CLINICAL TRIAL: NCT04598347
Title: Valuation of the Possible Vertical Transmission of SARS-CoV-2 Through Study of Amniotic Fluid and Chorionic Villi of Affected Pregnant Women for the COVID-19
Brief Title: Evaluation of the Possible Vertical Transmission of SARS-CoV-2 Through Study of Amniotic Fluid and Chorionic Villi of Affected Pregnant Women for the COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2020-59
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Pregnancy Related
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — umbilical cord blood, samples from the neonatal nasopharynx, the amnio-chorion interface, and placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women diagnosed with SARS-CoV-2: Pregnant women diagnosed with SARS-CoV-2 infection(by PCR on nasopharyngeal aspirate or serology)that have an indication to perform an invasive technique(chorionic biopsy or amniocentesis) along thegestation.The sample size will depend on the duration of theSARS-CoV-2 pandemic.Initially we propose a study period of 18months in which we would have an approximate total of 225pregnant women with indication of invasive technique.It is planned to conduct a PCR study for SARS-CoV-2 in amniotic fluid or chorionic villi to thosepregnant women diagnosed with SARS-CoV-2 infection(approximately 5% of the total pregnant womenwith indication of invasive technique (11-12 pregnant women)).This determination is made as part of theroutine clinical practice in the context of the study of screening for perinatal infections

SUMMARY:
Longitudinal prospective study in pregnant women withpositive serology or PCR for SARS-CoV-2 and indicationinvasive technique (amniocentesis or chorionic biopsy) that has the objective to evaluate the possible vertical transmission of SARS-CoV-2in the amniotic fluid or chorionic villi of pregnant women affected by coronavirus in the different periods of gestation.

DETAILED DESCRIPTION:
Patients will be recruited at the time theypresent an indication to perform a techniqueinvasive (amniocentesis or chorion biopsy). Eitherscreening for first or second trimester aneuploidies ofhigh risk, due to the presence of fetal malformation, due toearly intrauterine growth retardation (ICR) or due tosuspected chorioamnionitis.

The study population will be pregnant women diagnosed with SARS-CoV-2 infection(by PCR on nasopharyngeal aspirate or serology)that have an indication to perform an invasive technique(chorionic biopsy or amniocentesis) along thegestation.The sample size will depend on the duration of theSARS-CoV-2 pandemic.Initially we propose a study period of 18 months in which we would have an approximate total of 225 pregnant women with indication of invasive technique.It is planned to conduct a PCR study for SARS-CoV-2 in amniotic fluid or chorionic villi to those pregnant women diagnosed with SARS-CoV-2 infection(approximately 5% of the total pregnant womenwith indication of invasive technique (11-12 pregnant women)).This determination is made as part of theroutine clinical practice in the context of the study ofscreening for perinatal infections.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with SARS-CoV-2 (by PCR in aspiratenasopharyngeal or serologies)
* Patients indicated for an invasive technique(chorionic biopsy or amniocentesis

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: regnant women diagnosed with SARS-CoV-2 (by PCR in aspiratenasopharyngeal or serologies) that indicate an invasive technique(chorionic biopsy or amniocentesis) throughout pregnancy either due to high riskof aneuploidies in the first or second trimester screening, due to the presence offetal malformation, due to diagnosis of early intrauterine growth retardation (ICR)or for suspected chorioamnionitis.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2022-01-08 (Estimated); Study Completion 2022-01-23 (Estimated)

PRIMARY OUTCOMES:
Perinatal SARS-CoV-2 infection | 15 days
  Presence of SARS-CoV-2 in amniotic fluid or villichorionics from pregnant women with positive serology or PCR in nasopharyngeal aspirate duringgestation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
A specific database will be created for the study in which each patient will beAnonymously encoded in such a way that it is not identifiable.The person responsible for database creation, data entry and analysisstatistician will be Dra. Obdulia Alejos Abad.

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Breslin N, Baptiste C, Gyamfi-Bannerman C, Miller R, Martinez R, Bernstein K, Ring L, Landau R, Purisch S, Friedman AM, Fuchs K, Sutton D, Andrikopoulou M, Rupley D, Sheen JJ, Aubey J, Zork N, Moroz L, Mourad M, Wapner R, Simpson LL, D'Alton ME, Goffman D. Coronavirus disease 2019 infection among asymptomatic and symptomatic pregnant women: two weeks of confirmed presentations to an affiliated pair of New York City hospitals. Am J Obstet Gynecol MFM. 2020 May;2(2):100118. doi: 10.1016/j.ajogmf.2020.100118. Epub 2020 Apr 9. PMID 32292903
- [Background] Garg S, Kim L, Whitaker M, O'Halloran A, Cummings C, Holstein R, Prill M, Chai SJ, Kirley PD, Alden NB, Kawasaki B, Yousey-Hindes K, Niccolai L, Anderson EJ, Openo KP, Weigel A, Monroe ML, Ryan P, Henderson J, Kim S, Como-Sabetti K, Lynfield R, Sosin D, Torres S, Muse A, Bennett NM, Billing L, Sutton M, West N, Schaffner W, Talbot HK, Aquino C, George A, Budd A, Brammer L, Langley G, Hall AJ, Fry A. Hospitalization Rates and Characteristics of Patients Hospitalized with Laboratory-Confirmed Coronavirus Disease 2019 - COVID-NET, 14 States, March 1-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):458-464. doi: 10.15585/mmwr.mm6915e3. PMID 32298251
- [Background] Di Mascio D, Khalil A, Saccone G, Rizzo G, Buca D, Liberati M, Vecchiet J, Nappi L, Scambia G, Berghella V, D'Antonio F. Outcome of coronavirus spectrum infections (SARS, MERS, COVID-19) during pregnancy: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2020 May;2(2):100107. doi: 10.1016/j.ajogmf.2020.100107. Epub 2020 Mar 25. PMID 32292902
- [Background] Schwartz DA. An Analysis of 38 Pregnant Women With COVID-19, Their Newborn Infants, and Maternal-Fetal Transmission of SARS-CoV-2: Maternal Coronavirus Infections and Pregnancy Outcomes. Arch Pathol Lab Med. 2020 Jul 1;144(7):799-805. doi: 10.5858/arpa.2020-0901-SA. PMID 32180426
- [Background] Khan S, Jun L, Nawsherwan, Siddique R, Li Y, Han G, Xue M, Nabi G, Liu J. Association of COVID-19 with pregnancy outcomes in health-care workers and general women. Clin Microbiol Infect. 2020 Jun;26(6):788-790. doi: 10.1016/j.cmi.2020.03.034. Epub 2020 Apr 8. No abstract available. PMID 32278081
- [Background] Sutton D, Fuchs K, D'Alton M, Goffman D. Universal Screening for SARS-CoV-2 in Women Admitted for Delivery. N Engl J Med. 2020 May 28;382(22):2163-2164. doi: 10.1056/NEJMc2009316. Epub 2020 Apr 13. No abstract available. PMID 32283004
- [Background] Della Gatta AN, Rizzo R, Pilu G, Simonazzi G. Coronavirus disease 2019 during pregnancy: a systematic review of reported cases. Am J Obstet Gynecol. 2020 Jul;223(1):36-41. doi: 10.1016/j.ajog.2020.04.013. Epub 2020 Apr 18. PMID 32311350
- [Background] Qiancheng X, Jian S, Lingling P, Lei H, Xiaogan J, Weihua L, Gang Y, Shirong L, Zhen W, GuoPing X, Lei Z; sixth batch of Anhui medical team aiding Wuhan for COVID-19. Coronavirus disease 2019 in pregnancy. Int J Infect Dis. 2020 Jun;95:376-383. doi: 10.1016/j.ijid.2020.04.065. Epub 2020 Apr 27. PMID 32353549
- [Background] Yang Z, Wang M, Zhu Z, Liu Y. Coronavirus disease 2019 (COVID-19) and pregnancy: a systematic review. J Matern Fetal Neonatal Med. 2022 Apr;35(8):1619-1622. doi: 10.1080/14767058.2020.1759541. Epub 2020 Apr 30. PMID 32354293
- [Background] Li N, Han L, Peng M, Lv Y, Ouyang Y, Liu K, Yue L, Li Q, Sun G, Chen L, Yang L. Maternal and Neonatal Outcomes of Pregnant Women With Coronavirus Disease 2019 (COVID-19) Pneumonia: A Case-Control Study. Clin Infect Dis. 2020 Nov 19;71(16):2035-2041. doi: 10.1093/cid/ciaa352. PMID 32249918
- [Background] CDC COVID-19 Response Team. Preliminary Estimates of the Prevalence of Selected Underlying Health Conditions Among Patients with Coronavirus Disease 2019 - United States, February 12-March 28, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):382-386. doi: 10.15585/mmwr.mm6913e2. PMID 32240123
- [Background] Mullins E, Evans D, Viner RM, O'Brien P, Morris E. Coronavirus in pregnancy and delivery: rapid review. Ultrasound Obstet Gynecol. 2020 May;55(5):586-592. doi: 10.1002/uog.22014. PMID 32180292
- [Background] Karami P, Naghavi M, Feyzi A, Aghamohammadi M, Novin MS, Mobaien A, Qorbanisani M, Karami A, Norooznezhad AH. WITHDRAWN: Mortality of a pregnant patient diagnosed with COVID-19: A case report with clinical, radiological, and histopathological findings. Travel Med Infect Dis. 2020 Apr 11:101665. doi: 10.1016/j.tmaid.2020.101665. Online ahead of print. No abstract available. PMID 32283217
- [Background] Hantoushzadeh S, Shamshirsaz AA, Aleyasin A, Seferovic MD, Aski SK, Arian SE, Pooransari P, Ghotbizadeh F, Aalipour S, Soleimani Z, Naemi M, Molaei B, Ahangari R, Salehi M, Oskoei AD, Pirozan P, Darkhaneh RF, Laki MG, Farani AK, Atrak S, Miri MM, Kouchek M, Shojaei S, Hadavand F, Keikha F, Hosseini MS, Borna S, Ariana S, Shariat M, Fatemi A, Nouri B, Nekooghadam SM, Aagaard K. Maternal death due to COVID-19. Am J Obstet Gynecol. 2020 Jul;223(1):109.e1-109.e16. doi: 10.1016/j.ajog.2020.04.030. Epub 2020 Apr 28. PMID 32360108
- [Background] Elshafeey F, Magdi R, Hindi N, Elshebiny M, Farrag N, Mahdy S, Sabbour M, Gebril S, Nasser M, Kamel M, Amir A, Maher Emara M, Nabhan A. A systematic scoping review of COVID-19 during pregnancy and childbirth. Int J Gynaecol Obstet. 2020 Jul;150(1):47-52. doi: 10.1002/ijgo.13182. Epub 2020 May 17. PMID 32330287
- [Background] Yan J, Guo J, Fan C, Juan J, Yu X, Li J, Feng L, Li C, Chen H, Qiao Y, Lei D, Wang C, Xiong G, Xiao F, He W, Pang Q, Hu X, Wang S, Chen D, Zhang Y, Poon LC, Yang H. Coronavirus disease 2019 in pregnant women: a report based on 116 cases. Am J Obstet Gynecol. 2020 Jul;223(1):111.e1-111.e14. doi: 10.1016/j.ajog.2020.04.014. Epub 2020 Apr 23. PMID 32335053
- [Background] Li J, Wang Y, Zeng Y, Song T, Pan X, Jia M, He F, Hou L, Li B, He S, Chen D. Critically ill pregnant patient with COVID-19 and neonatal death within two hours of birth. Int J Gynaecol Obstet. 2020 Jul;150(1):126-128. doi: 10.1002/ijgo.13189. Epub 2020 May 27. PMID 32369616
- [Background] Qiu L, Liu X, Xiao M, Xie J, Cao W, Liu Z, Morse A, Xie Y, Li T, Zhu L. SARS-CoV-2 Is Not Detectable in the Vaginal Fluid of Women With Severe COVID-19 Infection. Clin Infect Dis. 2020 Jul 28;71(15):813-817. doi: 10.1093/cid/ciaa375. PMID 32241022
- [Background] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Background] Baud D, Greub G, Favre G, Gengler C, Jaton K, Dubruc E, Pomar L. Second-Trimester Miscarriage in a Pregnant Woman With SARS-CoV-2 Infection. JAMA. 2020 Jun 2;323(21):2198-2200. doi: 10.1001/jama.2020.7233. PMID 32352491
- [Background] Penfield CA, Brubaker SG, Limaye MA, Lighter J, Ratner AJ, Thomas KM, Meyer JA, Roman AS. Detection of severe acute respiratory syndrome coronavirus 2 in placental and fetal membrane samples. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100133. doi: 10.1016/j.ajogmf.2020.100133. Epub 2020 May 8. No abstract available. PMID 32391518
- [Background] Dong L, Tian J, He S, Zhu C, Wang J, Liu C, Yang J. Possible Vertical Transmission of SARS-CoV-2 From an Infected Mother to Her Newborn. JAMA. 2020 May 12;323(18):1846-1848. doi: 10.1001/jama.2020.4621. PMID 32215581
- [Background] Alzamora MC, Paredes T, Caceres D, Webb CM, Valdez LM, La Rosa M. Severe COVID-19 during Pregnancy and Possible Vertical Transmission. Am J Perinatol. 2020 Jun;37(8):861-865. doi: 10.1055/s-0040-1710050. Epub 2020 Apr 18. PMID 32305046
- [Background] Kimberlin DW, Stagno S. Can SARS-CoV-2 Infection Be Acquired In Utero?: More Definitive Evidence Is Needed. JAMA. 2020 May 12;323(18):1788-1789. doi: 10.1001/jama.2020.4868. No abstract available. PMID 32215579